CLINICAL TRIAL: NCT02010866
Title: Reaching Out to Distressed Medical Residents, Fellows, and Faculty Through the OHSU Resident and Faculty Wellness Program Interactive Screening Program (ISP)
Brief Title: Reaching Out to Distressed Medical Residents, Fellows and Faculty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Marie Soller, Professor, Psychiatry, Resident and Faculty Wellness, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 00009003
Record Dates: First submitted 2013-11-27; First posted 2013-12-13 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Depression; Suicide
Keywords: internship and residency; physicians; prevention; counseling; suicide; depression; burnout
MeSH Terms: conditions — Depression; Suicide; Burnout, Psychological | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Counseling (Other): in-person counseling through RFWP to distressed respondents on the ISP and patients who seek counseling without completing the ISP
  Interventions: Behavioral: counseling

INTERVENTIONS:
Behavioral: counseling — in-person counseling through RFWP offered to distressed respondents on the ISP and others who seek counseling (due to other reasons for referral)

SUMMARY:
The purpose of this study is to study whether distressed medical residents, fellows, and faculty health professionals benefit from completing online an anonymous and interactive screening of stress, depression, substance use, and suicidal thoughts. The screening and ability to interact online with a clinician anonymously are hypothesized to increase willingness to come for counseling in person. Suicide risk factors are expected to be lower once the distressed medical trainee or faculty member receives treatment.

DETAILED DESCRIPTION:
According to theories such as motivational interviewing and stages of change, individuals change health behaviors when the benefits (e.g., being less stressed) outweigh the risks (e.g., concerns about confidentiality of treatment). Prior research suggests that educational programming to promote the benefits and counter the perceived risks of counseling increases adults' motivation to get professional help. Distressed physicians' motivation to seek help following an educational intervention has not been evaluated but organizations such as the American Foundation for Suicide Prevention, Association for the Accreditation of Graduate Medical Education, and the American Medical Association have developed policies and programming to educate physicians about the importance of treating depression and reducing suicide risk in themselves and their colleagues.

A "best practices" suicide prevention program in 50+ US universities, the American Foundation for Suicide Prevention's Interactive Screening Program (ISP), was identified by the Oregon Health and Science University (OHSU) Resident and Faculty Wellness Program (RFWP) clinicians as a possible avenue by which to reach distressed OHSU trainees and faculty and encourage them to get help. The "Stress and Depression Questionnaire" is an anonymous, online screening tool for stress, depression, substance abuse, eating disorders, and suicide risk. Responses are scored and ranked according to level of distress and risk with Tier 1 representing "high risk, high distress" and Tier 2 "moderate distress, less risk" and Tier 3 "low or no distress or risk". RFWP clinicians will monitor responses, provide prompt communication back to the participants with information about how they scored, resources available to them, address any questions/concerns they might have and invite them to set up an appointment at the RFWP (if distressed). Moutier and her colleagues at a similar size academic medical center to OHSU, University of California at San Diego (UCSD), administered this survey to all medical students, residents, fellows, and faculty (13% completed it) and the majority eventually seen by clinicians indicated that they never would have sought help if they had not received feedback on the ISP and been encouraged to come in for evaluation/treatment. Being able to anonymously dialogue with a clinician about their specific situation and questions appeared to persuade some participants to come in for an evaluation or accept a referral. This academic medical center did not have an in-house counseling program for residents and faculty like the OHSU RFWP-UCSD trainees received an initial evaluation from a clinician and then were provided with community referrals. Their participation rate of 13% is similar to rates of participation in the ISP in undergraduate populations. In the present study, it is hypothesized that a highly visible and utilized RFWP may lead to a higher ISP participation rate among the residents, fellows, and faculty.

Although the ultimate goal is to save lives (i.e., reduce the rate of suicide among medical trainees and faculty), the low base rate of suicide in a population makes it difficult to evaluate whether the implementation of the ISP at OHSU will lead to a drop in suicide rates at this institution. Even using patient suicidal ideation and attempts as outcomes is problematic as this information can be difficult to gather unless the patient is actively involved in treatment at the time. Rather in the present study the effectiveness of this suicide prevention program will be measured by examining related variables to suicide risk-increases in protective factors and decreases in risk factors. Specifically, these researchers seek to decrease known risk factors (e.g., identify and intervene with untreated depression, substance abuse, high level of stress) and increase protective factors (e.g., promote self-awareness, receipt of support and resources and delivery of mental health services if needed).

Present study aims are to:

* reduce known risk factors of untreated psychological distress (e.g., depression, high stress level, substance abuse) by encouraging all residents, fellows, and School of Medicine (SOM) faculty to complete a self-assessment of their level of stress and risk using the ISP and then offer professional help through a personalized message/dialogue that directly addresses any concerns/barriers about seeking help at the RFWP and offers resources for better coping;
* increase self-awareness in mildly/moderately distressed trainees and faculty who fill out the ISP and offer preventive/early intervention educational resources via the ISP on topics that are relevant to them (based on their responses);
* evaluate whether all RFWP patients (ones who come to the program via ISP and other referral sources) report decreased psychological distress, burnout, and risk of suicide across treatment;
* assess levels of distress and flourishing among RFWP participants over time
* assess level of satisfaction with the RFWP educational outreach workshops, consultation to department leaders (and referral of their trainees and/or faculty), and clinical services provided to distressed trainees and faculty.

ELIGIBILITY:
Inclusion Criteria:

* OHSU medical residents, fellows, and full-time School of Medicine faculty

Exclusion Criteria:

* individuals not meeting the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
ISP levels of distress seen with medical trainees and faculty | Time survey is completed by trainee or faculty member at baseline
  online, anonymous Interactive Screening Program (ISP) measures stress, depression, anxiety, substance abuse, and suicidal ideation--participants fill out survey at different points and may or may not come in for counseling
Demographics of residents and faculty physicians who seek counseling through in house program | at enrollment for treatment (intake appointment)
  Demographics of residents, faculty at time of intake for counseling at Resident and Faculty Wellness Program
Who responds to treatment--level of distress | time of intake (baseline) to participants' end of treatment or 6 months since last seen
  % of participants in counseling services through Resident and Faculty Wellness who show change in psychological distress on ACORN from baseline to end of treatment
Who responds to treatment-level of burnout | time of intake to participants' end of treatment or 6 months since last seen
  participants at Resident and Faculty Wellness Program who show significant decline in burnout on MBI screening items (emotional exhaustion and depersonalization items) from baseline (time of intake) to end of treatment
Who responds to treatment-clinician rating of suicide risk | time of intake (baseline) to participants end of treatment or 6 months since last seen
  participants of Resident and Faculty Wellness Program who show change in clinician rating of suicide risk during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marie V Soller, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
will not be sharing data with other researchers outside of this project

DOCUMENTS (1):
  • Study Protocol (2024-04-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT02010866/Prot_000.pdf